CLINICAL TRIAL: NCT05744505
Title: 1565nm Non-ablative Fractional Laser Treat Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0797
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; 1565nm Non-ablative Fractional Laser; immune privilege
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): Every 3 weeks, a fixed 1 / 2 of the alopecia area was treated with a 1565-nm non-ablative fractional laser.
  Interventions: Procedure: 1565nm Non-ablative Fractional Laser
- control group (Placebo Comparator): There was no treatment for the other half of the alopecia area in the patients.
  Interventions: Procedure: placebo

INTERVENTIONS:
Procedure: 1565nm Non-ablative Fractional Laser — Every 3 weeks
  Arms: Laser group
Procedure: placebo — Every 3 weeks
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate and explore the mechanism of 1565-nm non-ablative fractional laser in the treatment of alopecia areata. The main questions it aims to answer are: (a) comparing the secretion of various cells and cytokines around and within hair follicles before and after treatment; (b) determining the Lord Want effector cells with cytokines and demonstrating that they mediate involvement in correcting the immune immunity collapse process. Participants' 1/2 of the treated alopecia area was compared to their own other half of the untreated alopecia area, and they were followed every three months for efficacy assessment and scalp biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years and ≤ 55 years of age;
* Alopecia areata subjects, and diagnosed with alopecia areata for 6 -12 months before screening;
* Women of childbearing age, non-pregnant or lactating, and subjects and their partners voluntarily take contraceptive measures deemed effective by the investigator during treatment and for at least 6 months after the last trial;
* Those who have no contraindications to the use of materials;
* Subject is able to understand and voluntarily sign the written informed consent form, which must be signed prior to the execution of any trial-specified study procedures;
* Subjects must be voluntary and able to complete the study procedure and follow-up examination.

Exclusion Criteria:

* Subjects who meet the diagnostic criteria for alopecia areata but are accompanied by the following diseases cannot be enrolled: local infection (bacterial, fungal or viral) at the site requiring laser treatment; Have a psychiatric disorder (e.g., schizophrenia, neurosis, organic psychosis, etc.);
* Subjects who have previously treated drugs or surgeries and cannot be enrolled in the following situations: receiving other anti-alopecia areata treatments (including topical glucocorticoids,microneedling, laser treatment, etc.) at the same time; Receiving any other clinical investigational drug treatment concurrently;
* Any other situation or condition in which the investigator considers that the subject is not suitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline alopecia area at one year | baseline and 3, 9, 12 months after the first treatment
  The range of alopecia area in patients receiving 1565nm Non-ablative Fractional Laser treatment was assessed by the hair loss severity scoring tool (SALT) to evaluate the efficacy every three months. The higher the score, the more severe the hair loss and the less effective the treatment.
Change from Baseline scalp biopsy at one week after the second laser treatment | baseline and one week after the second laser treatment
  Single-cell sequencing will be used to analyze CD8 + NKG 2 D + T cells, Th 1, Th 2, Th 17, and Treg cells before and after treatment, analyzing differences in cytokine secretion.

CONTACTS AND LOCATIONS:
Locations (1):
- Xianjie Wu, Hangzhou, Zhejiang, China